CLINICAL TRIAL: NCT05834127
Title: Comparative Effects of Aerobic Exercises and Yoga on Pain and Symptoms Severity in Premenstrual Syndrome
Brief Title: Effects of Aerobic Exercises and Yoga on Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0508
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Premenstrual Syndrome; Pain
Keywords: Aerobic exercises; Menstruation; Premenstrual syndrome; Visual analogue scale; Yoga
MeSH Terms: conditions — Premenstrual Syndrome; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercises (Experimental): Group A will receive aerobic exercises. Treatment will be given 3 times a week for 1 month. Total number of sessions will be 12
  Interventions: Other: Aerobic exercise
- Yoga exercises (Active Comparator): Group B will receive yoga. Treatment will be given for 40 min, 3 times a week for 1 month.
  Total number of sessions will be 12
  Interventions: Other: Yoga Exercises

INTERVENTIONS:
Other: Aerobic exercise — Group A will receive aerobic exercise in the form of warm up and cool down (both for 5 min)
  * Treadmill (30 min) based on Target Heart Rate (calculated using Karvina formula at 60%-70% of heart rate reserve).
  * Treatment will be given 3 times a week for 1 month
  Arms: Aerobic exercises
Other: Yoga Exercises — Group B will receive yoga movements for 40 min, 3 times a week for 1 month.
  * They will be given yoga movements, including 10 min of Kapalbharti Pranayama which includes automatic inhalation with short and forceful exhalations.
  * 20 min of yoga movements (Cat-cow pose, Child's pose, Plank pose, Cobra pose - each for 5 min).
  * 10 min of meditation/relaxation in Savasana pose
  Arms: Yoga exercises

SUMMARY:
Sign and symptoms including mood swings, sensitive breasts, food cravings, exhaustion, irritability, pain and sadness. The physical and emotional changes you go through with premenstrual syndrome can range from hardly perceptible to severe. Some people's physical discomfort and emotional stress are so severe that it interferes with their daily life. Regardless of the severity of the symptoms, most women's signs and symptoms go away four days following the start of their menstrual cycle. In this study the effects of aerobic exercises and Yoga on premenstrual syndrome population will be analyzed. This study will be a randomized clinical trial which will incorporate two different interventions. Aerobic exercises and yoga would be administered to the females. 32 patients will randomly divided into two groups. Assessment will be done by using PMS scale and visual analogue scale. The goal of this study to compare the effects of aerobic exercises and yoga on premenstrual syndrome.

DETAILED DESCRIPTION:
There are many different signs and symptoms of premenstrual syndrome (PMS), including mood swings, sensitive breasts, food cravings, exhaustion, irritability, pain and sadness. Premenstrual syndrome is thought to have affected up to 3 out of every 4 women who are menstruation. A consistent pattern of recurrence exists for symptoms. However, the physical and emotional changes you go through with premenstrual syndrome can range from hardly perceptible to severe. Some people's physical discomfort and emotional stress are so severe that it interferes with their daily life. Regardless of the severity of the symptoms, most women's signs and symptoms go away four days following the start of their menstrual cycle.

Various treatment options are available in the literature to effectively manage these issues through Pharmacotherapies. All these interventions are reported to have beneficial effect for these problems. In this study the effects of aerobic exercises and Yoga on premenstrual syndrome population will be analyzed. This study will be a randomized clinical trial which will incorporate two different interventions. Aerobic exercises and yoga would be administered to the females. 32 patients will randomly divided into two groups. Assessment will be done by using PMS scale and visual analogue scale. The goal of this study to compare the effects of aerobic exercises and yoga on premenstrual syndrome. Subjects meeting the predetermined inclusion criteria will be divided into two groups. 1stgroup will be treated with aerobic exercise. 2nd group will be treated with yoga movements. The pain intensity (Visual Analog Scale) and PMS Scale will be measured before, at the end of 15 days, and after 1 month of treatment program. Recorded values will be analyzed for any change using SPSS25.

ELIGIBILITY:
Inclusion Criteria

* Age between 16 and 45 years
* No history of any mental and physical diseases
* No history of joint, motion, muscle, and bone diseases that reduce their abilities of exercise
* Not on any medication and mineral supplements during three menstrual cycles
* Having regular menstrual cycles 24 to 35 days
* No incidents such as relatives' death, marriage, or any medical emergency in the last 3 months

Exclusion Criteria

* Not able to tolerate physical exercise
* Any history of gynecological surgery
* Professional athletes
* Chronic disease: diabetes, hypertension, cardiac disease, infectious disease
* Irregular and infrequent menstrual cycle
* Using intrauterine devices and hormonal therapy
* Pregnant Females

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Because PMS condition is only present in females
Enrollment: 36 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 4 weeks
  Operationally a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end, as illustrated. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks
PMS Scale(premenstrual syndrome scale) | 4 weeks
  Premenstrual Syndrome Scale (PSS) was used based on Diagnostic and Statistical Manual III (DSM-III) and IV (revised)(DSM IV-R) for the evaluation of PMS. The scale consists of 44 items, 5 of which are Likert type. The scores range between 44 and 220 and those with a score of 133 and above are considered to have PMS

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, M.phil, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] A DM, K S, A D, Sattar K. Epidemiology of Premenstrual Syndrome (PMS)-A Systematic Review and Meta-Analysis Study. J Clin Diagn Res. 2014 Feb;8(2):106-9. doi: 10.7860/JCDR/2014/8024.4021. Epub 2014 Feb 3. PMID 24701496
- [Background] Derman O, Kanbur NO, Tokur TE, Kutluk T. Premenstrual syndrome and associated symptoms in adolescent girls. Eur J Obstet Gynecol Reprod Biol. 2004 Oct 15;116(2):201-6. doi: 10.1016/j.ejogrb.2004.04.021. PMID 15358465
- [Background] Steiner M, Steinberg S, Stewart D, Carter D, Berger C, Reid R, Grover D, Streiner D. Fluoxetine in the treatment of premenstrual dysphoria. Canadian Fluoxetine/Premenstrual Dysphoria Collaborative Study Group. N Engl J Med. 1995 Jun 8;332(23):1529-34. doi: 10.1056/NEJM199506083322301. PMID 7739706
- [Background] Chen KM, Tseng WS, Ting LF, Huang GF. Development and evaluation of a yoga exercise programme for older adults. J Adv Nurs. 2007 Feb;57(4):432-41. doi: 10.1111/j.1365-2648.2007.04115.x. PMID 17291207
- [Background] Vaghela N, Mishra D, Sheth M, Dani VB. To compare the effects of aerobic exercise and yoga on Premenstrual syndrome. J Educ Health Promot. 2019 Oct 24;8:199. doi: 10.4103/jehp.jehp_50_19. eCollection 2019. PMID 31867375
- [Background] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679
- [Background] Ghaffarilaleh G, Ghaffarilaleh V, Sanamno Z, Kamalifard M, Alibaf L. Effects of Yoga on Quality of Sleep of Women With Premenstrual Syndrome. Altern Ther Health Med. 2019 Sep;25(5):40-47. PMID 31221931